CLINICAL TRIAL: NCT01207076
Title: Phase I Open Label, Single Arm, Dose Escalation Trial to Evaluate the Biodistribution and Safety of AHN-12 In Patients With Advanced Leukemia HM2010-05
Brief Title: AHN-12 Biodistribution in Advanced Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010LS030
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia
Keywords: CD45+ disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- receiving AHN-12 and 90Y-AHN-12 (Experimental): Patients receiving nonradiolabeled cold AHN-12 (.20 mg/kg to 1.0 mg/kg) of at least one dose and up to a total of 3 dosimetry infusions (intervals no sooner than 8 days and up to 21 days).
  Interventions: Biological: 90Y-AHN-12

INTERVENTIONS:
Biological: 90Y-AHN-12 — The intervention consists of two parts.
  1. The dose of cold AHN-12 to achieve favorable biodistribution through imaging using 111In-AHN-12.
     * Dose escalation of nonradiolabeled AHN-12:
     Dose level= -1 0.20 mg/kg, Dose level=1 0.40 mg/kg, Dose level=2 0.80 mg/kg, Dose level=3 1.20 mg/kg, Dose level=4 1.60 mg/kg, Dose level=5 2.00 mg/kg
  2. Phase I therapeutic dosing of cold AHN-12 at dose established plus 90Y-AHN-12.
     * the starting 90Y-AHN-12 dose level will be 4 Gy with the dose escalated in increments of 4 Gy to a maximum of 20 Gy.

SUMMARY:
This study is a single institution phase I study for the treatment of patients with relapsed or refractory leukemia aged 12 years and older using 90Y-AHN-12.

DETAILED DESCRIPTION:
A dose escalation schema will be used with the initial patient receiving the current lowest dose of nonradiolabeled AHN-12 (from 0.20 mg/kg to 1.0 mg/kg). If a favorable biodistribution is not achieved and the patient remains negative for HAMA, the infusion may be repeated up to two more times (with a one level increase in nonradiolabeled AHN-12 each time) in an attempt of achieving favorable biodistribution.

In order to achieve the primary objective of identifying the optimal nonradiolabeled dose of AHN-12 antibody for all patients, if the first patient at the current antibody dose does not achieve favorable biodistribution, the next patient(s) will be treated at the next higher dose level.

Patients achieving favorable biodistribution and remaining negative for HAMA will be eligible for the therapeutic component of this trial. Those not meeting these requirements will be taken off study and followed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following histologically confirmed CD45+ diseases. If possible, AHN-12 positivity will be confirmed by flow cytometry on a recent bone marrow or a peripheral blood sample, if circulating blasts are present.

  * Acute myelogenous leukemia (AML), primary refractory or relapsed disease
  * Refractory myelodysplastic syndrome (MDS)
  * AML arising from pre-existing MDS, refractory
  * Acute lymphoblastic leukemia (ALL), primary refractory or relapsed disease
  * Chronic myelogenous leukemia (CML) following blast crisis
* Age ≥ 12 years
* Karnofsky Performance Status ≥ 60% (16 years and older) or Lansky Play Score ≥ 60 (<16 years)
* Life expectancy of > 12 weeks in the opinion of the enrolling medical provider
* Patients must have adequate organ function
* Human anti-mouse antibody (HAMA) must be negative (perform on all patients regardless of prior therapies).
* Consent to adequate contraception. The effects of 90Y-AHN-12 on the developing fetus are unknown.
* Source of allogeneic stem cells must have been identified in event of severe myelosuppression
* Able to give written consent.
* Both men and women of all ethnic groups are eligible for this trial.

Exclusion Criteria:

* Ongoing grade 2 or greater non-hematologic toxicity due to previously administered therapies
* < 8 days from completion of therapy with any biologic agent
* Receiving any investigational agents
* Active central nervous system (CNS) leukemia are excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 90Y-AHN-12 or other agents used in study.
* Uncontrolled illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the enrolling medical provider.
* Pregnant and breastfeeding women are excluded from this study because 90Y-AHN-12, being radioactive, as well as high dose chemotherapy and total body irradiation (TBI) have the potential for teratogenic or abortifacient effects.
* Human immunodeficiency virus (HIV) positive patients:
* < 60 days since an autologous transplant
* Bone marrow cellularity <5% (because of concern of myelosuppression)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Optimal Dose of AHN-12 Non-radiolabeled Antibody | Day 2
  doses of nonradiolabeled antibody are specified: 0.20, 0.40, 0.60, 0.80 and 1.00 mg/kg.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of 90Y-AHN-12 | Within 14 days of achieving favorable biodistribution
  •Determine the MTD of 90Y-AHN-12 for patients with a favorable biodistribution and a negative human anti-mouse antibody (HAMA). Doses of radiolabeled antibody are specified starting dose level with dose increment of 2 gray (Gy) to maximum of 22 Gy.
Human Anti-Mouse Antibody (HAMA) Response | 30 and 90 Days Post Therapy, Then Every 6 Months If Positive
  Event is whether or not the patient develops a HAMA response.
Anti-tumor Activity of 90Y-AHN-12 | 30 and 90 Days Post Therapy
  Event is response to therapy: complete remission, partial remission, refractory or relapsed disease.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Burns, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States